CLINICAL TRIAL: NCT06420609
Title: Efficacy of a Proactive Approach to Death Thoughts in People with Advanced Cancer: a Randomized Clinical Trial
Brief Title: Efficacy of a Proactive Approach to Death Thoughts in People with Advanced Cancer
Acronym: Go-TAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Institut Català d'Oncologia (Other); Hospital Arnau de Vilanova (Other); Fundacion Rioja Salud (Other)
Responsible Party: Principal Investigator, Iris Crespo Martin, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PI22/01536
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Death; Advanced Cancer
MeSH Terms: conditions — Death

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study proposes a randomized controlled clinical trial (RCT) with a stepped-wedge design, in which 6 palliative care units from second and third level hospitals in Spain will collaborate. The six units will contribute with both experimental and control participants, starting with the recruitment of the control group participants and subsequently starting the intervention group. The time at which they will transition to the intervention will be chosen at random. The centers will be randomized to know at what point in the study they should begin the intervention and each center will be informed of the number of patients they should include in each of the groups. The clusters correspond to the different palliative care units that participate in the study. Six sequences will be carried out, seven periods with 4 patients in each period. Patients will be different in each of the periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Go-TAD (Experimental): the participants will receive a medical visit that will include the 4 open-ended questions comprising the Go-TAD intervention
  Interventions: Other: Go-TAD
- CONTROL (No Intervention): the participants will receive a medical visit that will include the 4 open-ended questions comprising hobbies and other personal themes, but not death.

INTERVENTIONS:
Other: Go-TAD — The participants will receive a medical visit that will include the 4 open-ended questions comprising the Go-TAD intervention
  Arms: Go-TAD

SUMMARY:
The aim of this study is to demonstrate the efficacy of a proactive intervention to approach death thoughts among people with advanced cancer compared to usual care (the reactive approach) via a feasible approach with previous indicators of efficacy: Go-TAD (Give the Opportunity to Talk about Death). The benefits of the intervention will be evaluated in terms of: reduction of emotional distress and hopelessness and improvement the doctor-patient relationship, as well as improvement of quality of life for the patient. A Phase II randomized controlled mixed methods clinical trial (RCT) will be carried out within 4 Palliative Care units of tertiary care hospitals in Catalonia. Participants will be persons with advanced cancer defined according to the criteria of the American Society of Clinical Oncology. Participants will be randomly assigned to an intervention group or control group. In the intervention group, the participants will receive a medical visit that will include the 4 open-ended questions comprising the Go-TAD intervention, while the control group will receive usual care. Between 24 and 96 hours later, a researcher from outside the center will assess study outcome measures. To strengthen the study conclusions, a qualitative study will be carried out in which the experiences of the participants in the intervention group and of their professionals who administered the Go-TAD will be explored in depth.

ELIGIBILITY:
The inclusion criteria will be:

1. patients with advanced cancer defined according to ASCO (American Society of Clinical Oncology) criteria referred for the initial palliative care (PC) consultation.
2. age over 18 years
3. ECOG 0-3 (functionality status)
4. outpatients and inpatients
5. patients who can sign the informed consent
6. patients with the ability to maintain a conversation

The exclusion criteria will be:

1. patients with acute symptoms that may affect their consciousness.
2. patients with any uncontrolled symptoms that prevent collaboration in the study assessed according to clinical judgment
3. moderate or severe cognitive impairment assessed according to clinical judgment
4. patients included in another incompatible clinical trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Emotional distress | 4 days
  The main outcome will be emotional distress, which will be evaluated using an instrument validated and developed in the context of palliative care in Spain, the Emotional Distress Detection (DME) questionnaire. This questionnaire is characterized by the simplicity and ease of application and the short application time, given that it only consists of 4 items. The first three items are questions with answers in the format of a visual numerical scale from 0 to 10, in which the state of mind and the perception of coping with the situation are evaluated, and another that records the presence or absence of concerns. The last question is based on the observation, by the healthcare professional, of the presence of external signs of emotional distress. The DME gives a total score (0 to 20) made up of the sum of the scores of the first three items, one of them in reverse format, with the highest scores indicating greater discomfort.

SECONDARY OUTCOMES:
Hopelessness assessed by the Beck Hopelessness Questionnaire (BHQ). | 4 days
  Hopelessness will be assessed with the Beck Hopelessness Questionnaire (BHQ). This validated and widely used questionnaire in palliative care research originally consists of 20 items that were reduced to 7 items with true/false responses in a brief version specially adapted to the area of palliative care. The total score ranges from 0 to 7, with higher scores indicating a higher level of hopelessness.
Doctor-patient relationship evaluated with the Patient-Doctor-Relationship Questionnaire -PDRQ-9-. | 4 days
  The quality of the doctor-patient relationship from the patient's perspective will be evaluated with the Patient-Doctor-Relationship Questionnaire -PDRQ-9-. This questionnaire consists of 9 items with a 5-point Likert-type response format and has been previously used in the field of palliative care. The total score ranges between 9-45, with higher scores indicating a better relationship between doctor and patient.
Quality of life related to health evaluated using the Palliative Outcome Scale (POS) | 4 days
  It will be evaluated using the Palliative Outcome Scale (POS). This scale has been validated with a proxy for quality of life in patients with palliative care. It consists of 12 items with multiple response format that address the physical and psychological dimensions, the information given, communication with family and friends, the meaning of life and other practical aspects related to the disease. The range of scores is 0-40, with higher scores indicating worse quality of life.

OTHER OUTCOMES:
Clinical and sociodemographic variables | 4 days
  age, gender, marital status, type of cancer, months since diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JJ, Liu DD. A predictive probability design for phase II cancer clinical trials. Clin Trials. 2008;5(2):93-106. doi: 10.1177/1740774508089279. PMID 18375647
- [Background] Limonero JT, Mateo D, Mate-Mendez J, Gonzalez-Barboteo J, Bayes R, Bernaus M, Casas C, Lopez M, Sirgo A, Viel S. [Assessment of the psychometric properties of the Detection of Emotional Distress Scale in cancer patients]. Gac Sanit. 2012 Mar-Apr;26(2):145-52. doi: 10.1016/j.gaceta.2011.07.016. Epub 2011 Oct 26. Spanish. PMID 22033008
- [Background] Martin-Fernandez J, del Cura-Gonzalez MI, Gomez-Gascon T, Fernandez-Lopez E, Pajares-Carabajal G, Moreno-Jimenez B. [Patient satisfaction with the patient-doctor relationship measured using the questionnaire (PDRQ-9)]. Aten Primaria. 2010 Apr;42(4):196-203. doi: 10.1016/j.aprim.2009.09.026. Epub 2010 Feb 8. Spanish. PMID 20116893
- [Background] Crespo I, Monforte-Royo C, Balaguer A, Pergolizzi D, Cruz-Sequeiros C, Luque-Blanco A, Porta-Sales J. Screening for the Desire to Die in the First Palliative Care Encounter: A Proof-of-Concept Study. J Palliat Med. 2021 Apr;24(4):570-573. doi: 10.1089/jpm.2020.0276. Epub 2020 Sep 18. PMID 32945714
- [Background] Serra-Prat M, Nabal M, Santacruz V, Picaza JM, Trelis J; Grupo Catalan de Estudio de la Efectividad de los Cuidados Paliativos. [Validation of the Spanish version of the Palliative Care Outcome Scale]. Med Clin (Barc). 2004 Oct 2;123(11):406-12. doi: 10.1016/s0025-7753(04)74535-2. Spanish. PMID 15482713
- [Background] Porta-Sales J, Crespo I, Monforte-Royo C, Marin M, Abenia-Chavarria S, Balaguer A. The clinical evaluation of the wish to hasten death is not upsetting for advanced cancer patients: A cross-sectional study. Palliat Med. 2019 Jun;33(6):570-577. doi: 10.1177/0269216318824526. Epub 2019 Jan 28. PMID 30688146
- [Derived] Julia-Torras J, Garcia-Salanova A, Monforte-Royo C, Jimeno Ariztia M, Balaguer A, Crespo I. Impact of proactively inviting people with advanced cancer to talk about the end of life: a randomised clinical trial protocol. BMJ Open. 2025 Jul 13;15(7):e104195. doi: 10.1136/bmjopen-2025-104195. PMID 40659391